CLINICAL TRIAL: NCT04187222
Title: Clinical Effect of Probiotic Use Bifidobacterium Animalis Subsp. Lactis as Adjunctive Therapy in Non-surgical Treatment of Periimplant Mucositis: a Randomized Controlled Trial
Brief Title: Effect of Probiotic Use Bifidobacterium Animalis Subsp. Lactis in Peri-implant Mucositis
Acronym: Mucosite prob
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Michel Reis Messora, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 82840117.4.0000.5419
Record Dates: First submitted 2019-11-25; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Mucositis Oral
Keywords: Dental implants; Mucositis; Probiotics; Bleeding on probing
MeSH Terms: conditions — Stomatitis; Mucositis

STUDY DESIGN:
Intervention Model Description: Treatment of peri-implant mucositis and maintenance care Prior to the beginning of the intervention, all patients received oral hygiene instruction. Mechanical debridements were performed with titanium curves and polishing using a rubber bowl and polishing paste. In the Test Group the treatment session was completed by a professional topical application around the carboxymethylcellulose gel implants containing 109 CFLs of B. lactis HN019. The gel was applied sub and supragingivally. The patients then received commercial capsules containing the same bacteria and were instructed to dissolve the capsule contents in 20 mL of water and rinse for 30 to 60 seconds, followed by swallowing twice a day for 12 weeks. The control group received the same oral hygiene instructions, mechanical debridement and was treated with gel and placebo tablets. At 3 months postoperatively, the same local mechanical and chemical treatment was repeated for the Test and Control groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Mechanical treatment + Bifidobacterium animalis subsp. lactis
  Interventions: Other: Mechanical debridements; Biological: Bifidobacterium animalis subsp. lactis
- Control Group (Placebo Comparator): Mechanical treatment + Placebo
  Interventions: Other: Mechanical debridements

INTERVENTIONS:
Other: Mechanical debridements — Prior to the beginning of the intervention, all patients received oral hygiene instruction. Mechanical debridements were performed with titanium curette and polishing using a rubber bowl and polishing paste.
Biological: Bifidobacterium animalis subsp. lactis — Capsules containing Bifidobacterium animalis subsp. lactis were chubby and subsequently ingested twice a day for 12 weeks.
  Arms: Test Group

SUMMARY:
Peri-implant disease is an inflammatory process of bacterial etiology that can affect the tissues around the implants and can be classified as peri-implant mucositis or peri-implantitis. The confirmation of the action of probiotics against microorganisms that cause peri-implant diseases can represent a great advance in the treatment of these diseases that affect a large part of the population, and may even reduce or prevent the use of antibiotics, reducing the risk of implant loss and, consequently, greater damage to the oral and systemic health of individuals. The purpose of this study was to evaluate the action of probiotics on the peri-implant health of total edentulous patients using Branemark protocol prosthetic rehabilitations. For this, 38 patients were selected, without systemic alterations and non-smokers. Clinical monitoring was performed at baseline (pre-intervention period) as well as at 12 and 24 weeks after study initiation. The following parameters were evaluated: modified gingival index (MGI), modified plaque index (MPI), probing depth (PD) and probing bleeding (PB). Data were subjected to statistical analysis at a significance level of 5%. There was an increase in sites with IGM 0 in the test group at 12 and 24 weeks. The test group presented more sites with IGM 0 than the control. IPM 0 sites increased in the control group at 12 and 24 weeks in the control group. PD decreases in a test and control group. Finally, the test group had lower PB rates. Thus, the probiotic used demonstrated ability to contribute to the improvement of peri-implant health of the patients analyzed.

DETAILED DESCRIPTION:
Clinical monitoring. MGI (0: no bleeding when a periodontal tube is passed along the mucosal margin adjacent to the implant; 1: visible isolated bleeding points; 2: blood forms a confluent red line at the mucosal margin and 3: profuse bleeding) and the MPI (0: no plaque; 1: plaque recognized only by probing through the smooth marginal surface of the implant; 2: plaque can be seen with the naked eye; 3: abundance of alba matter). PD was determined using a soft plastic periodontal probe for torque-controlled implants at 0.15 N / cm. Three buccal and three lingual reference points for each implant were used to calculate the mean probing depth in millimeters for each implant. PB was dichotomously evaluated: the presence of bleeding was considered positive when it occurred within 20 seconds after insertion of the probe to measure PD. The height of the keratinized mucosa present around each implant was also measured.

All clinical parameters described above were recorded at baseline (pre-intervention period) as well as at 12 and 24 weeks after study initiation.

Treatment of peri-implant mucositis and maintenance care. Prior to the beginning of the intervention, all patients received oral hygiene instruction. Mechanical debridements were performed with titanium curves and polishing using a rubber bowl and polishing paste. In the Test Group the treatment session was completed by a professional topical application around the carboxymethylcellulose gel implants containing 109 colony (CFU) forming units of B. lactis HN019. The gel was applied sub and supragingivally. The patients then received commercial capsules containing the same bacteria and were instructed to dissolve the capsule contents in 20 mL of water and rinse for 30 to 60 seconds, followed by swallowing twice a day for 12 weeks. The control group received the same oral hygiene instructions, mechanical debridement and was treated with gel and placebo tablets. At 3 months postoperatively, the same local mechanical and chemical treatment was repeated for the Test and Control groups.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous lower or upper dental arch undergoing rehabilitation with dental implants;
* prosthetic restoration in function for at least 6 months;
* healthy individuals with no known systemic changes;
* non smokers.

Exclusion Criteria:

* patients who have received any type of local or systemic oral cavity decontamination treatment within the last 3 months or periodontal treatment within the last 6 months; uncontrolled periodontal disease;
* patients with systemic disorders capable of influencing treatment outcomes;
* smokers;
* lack of informed consent to participate in the study;
* presence of bone loss greater than 2 mm in dental implants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Bleeding the probing. | Baseline.
Bleeding the probing. | 12 weeks.
Bleeding the probing. | 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry of Ribeirao Preto - University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Mongardini C, Pilloni A, Farina R, Di Tanna G, Zeza B. Adjunctive efficacy of probiotics in the treatment of experimental peri-implant mucositis with mechanical and photodynamic therapy: a randomized, cross-over clinical trial. J Clin Periodontol. 2017 Apr;44(4):410-417. doi: 10.1111/jcpe.12689. Epub 2017 Feb 18. PMID 28032908
- [Background] Hallstrom H, Lindgren S, Widen C, Renvert S, Twetman S. Probiotic supplements and debridement of peri-implant mucositis: a randomized controlled trial. Acta Odontol Scand. 2016;74(1):60-6. doi: 10.3109/00016357.2015.1040065. Epub 2015 May 8. PMID 25953193
- [Background] Flichy-Fernandez AJ, Ata-Ali J, Alegre-Domingo T, Candel-Marti E, Ata-Ali F, Palacio JR, Penarrocha-Diago M. The effect of orally administered probiotic Lactobacillus reuteri-containing tablets in peri-implant mucositis: a double-blind randomized controlled trial. J Periodontal Res. 2015 Dec;50(6):775-85. doi: 10.1111/jre.12264. Epub 2015 Feb 25. PMID 25712760
- [Derived] Santana SI, Silva PHF, Salvador SL, Casarin RCV, Furlaneto FAC, Messora MR. Adjuvant use of multispecies probiotic in the treatment of peri-implant mucositis: A randomized controlled trial. J Clin Periodontol. 2022 Aug;49(8):828-839. doi: 10.1111/jcpe.13663. Epub 2022 Jun 10. PMID 35634695